CLINICAL TRIAL: NCT00766064
Title: Effects of Paliperidone in Posttraumatic Stress Disorder (PTSD)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0804003717
Record Dates: First submitted 2008-09-30; First posted 2008-10-03 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone Dosing (Experimental): Paliperidone Dosing up to 6 weeks, with a maximum dosage of 6mg
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Paliperidone — Paliperidone will be gradually increased to a final dose between 3 - 6 mg/day according to the following schedule:
  Weeks 1 - 3: 3 mg daily, Weeks 4 - 5: flexible dosing according clinical situation, dose range between 3 mg - 6 mg daily*, Week 6: fixed dose,
  *Criteria to increase the dose from 3 mg to 6 mg daily are 1] absence of any side effects, 2] patients not showing a sufficient response to 3 mg paliperidone can be increased to 6 mg daily. Response is defined as change in depression and anxiety ratings of at least 30% compared to baseline.
  Other Names: Invega

SUMMARY:
Chronic posttraumatic stress disorder (PTSD) is a debilitating disorder and treatment response to pharmacological interventions has been modest for these patients. Chronic elevated anxiety and associated psychophysiological parameters including increased heart rate and alterations in skin conductance are key symptoms of chronic PTSD. Antidepressants, including selective serotonin reuptake inhibitors (SRIs) or norepinephrine-serotonin re-uptake inhibitors are considered treatment of first choice for these patients, however a substantial portion of patients do not respond sufficiently (Zhang and Davidson 2007). Therefore, there is a need to establish novel and effective add-on treatment strategies for these patients. Recently, atypical neuroleptics have received considerable attention since it was shown in multiple controlled and naturalistic trials that these medications are an effective treatment option for patients with PTSD (Davis et al 2006). In chronic PTSD, the psychophysiological responses at baseline and in response to treatment have yet been inadequately studied and may provide novel insight into antidepressant and anxiolytic mechanisms of medications used in the treatment of PTSD. Therefore, in addition to evaluating the antidepressant and anxiolytic effects of paliperidone, a novel atypical neuroleptic, in the treatment of PTSD, we also aim to compare neurophysiological responses at baseline with post-treatment effects in antidepressant-refractory PTSD patients.

Primary Aim 1: Evaluate the anxiolytic and antidepressant effects of paliperidone in patients with PTSD.

Secondary Aim 2: Evaluate the effects of paliperidone on fear conditioned psychophysiological responses (including startle eyeblink, skin conductance, and cardiovascular inter-beat interval) at baseline and after 6 weeks of naturalistic treatment in chronic PTSD patients.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in a naturalistic treatment study using paliperidone and in two fear conditioning tests, one at baseline and one at the end of the 6 weeks treatment study.
* We will include PTSD subjects on medications (possible medications include antidepressants, benzodiazepines) who have no or only partial treatment response. Paliperidone will be added to the existing treatment regime which will remain unchanged during the study period. PTSD subjects will have a minimum score of 50 on the Clinician-Administered PTSD Scale (CAPS; Blake et al, 1995).

Exclusion Criteria:

* a comorbid diagnosis of bipolar illness, schizophrenia or other psychotic disorders, acute or chronic suicidality, acute or chronic unstable medical conditions (including severely impaired hepatic function as indicated with abnormal PT and PTT, abnormal CBC, and liver enzymes more than 50% above the upper normal range, not well controlled blood pressure)
* current diagnosis of substance abuse or dependence
* unsuccessful treatment history with paliperidone
* known hypersensitivity to paliperidone or any of its inactive ingredients
* administration of any investigational drug up to 90 days before entry into the study
* intake of Class 1A (e.g., quinidine, procainamid) or Class III (e.g., amiodaronme, sotalol) antiarrhythmic medications, antipsychotics, antibiotics (e.g., gatifloxacin, moxifloxacin) (up to 90 days before entry into the study or during the study)
* subjects with a positive screen for drugs of abuse
* no startle or skin conductance response, or excessively high startle response to the startle probe (100 dB acoustic stimuli) during the pretest.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Behavioral ratings (e.g. MADRS, HAMA, CGI) and psychophysiological measures. Neurophysiological measurements of startle eyeblink, skin conductance, and cardiovascular inter-beat interval will be done. | behavioral ratings: weekly; Neurophysiological measurements will be done at baseline, before initiation of treatment with paliperidone (baseline) and after 6 weeks of paliperidone treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Neumeister, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States